CLINICAL TRIAL: NCT04120337
Title: Safe Access: Randomized Trial to Compare Removal Techniques for the One-Rod Subdermal Contraceptive Implant: RemovAid Device Versus Standard Approach
Brief Title: Safe Access: Trial With RemovAid Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RemovAid AS (Industry)
Collaborators: Karolinska Institutet (Other); Mulago Hospital, Uganda (Other); FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-103
Record Dates: First submitted 2019-10-01; First posted 2019-10-09 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-02

CONDITIONS: Removal of a Contraceptive Subdermal Implant
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RemovAid Device + lidocaine patch (Experimental): Test device with lidocaine patch for local anesthesia
  Interventions: Device: RemovAid device + lidocaine patch
- RemovAid Device + lidocaine injection (Experimental): Test device with lidocaine injection for local anesthesia
  Interventions: Device: RemovAid device + lidocaine injection
- Standard removal technique + lidocaine injection (Active Comparator): Standard technique involves a scalpel, forceps, and tweezers with lidocaine injection for local anesthesia
  Interventions: Procedure: Standard technique + lidocaine injection

INTERVENTIONS:
Device: RemovAid device + lidocaine patch — The RemovAid device incises the skin and grasps the implant for removal. A lidocaine patch will be used prior to incision.
  Arms: RemovAid Device + lidocaine patch
Procedure: Standard technique + lidocaine injection — Using scalpel, tweezers, and forceps to remove a subdermal implant. A lidocaine injection will be used prior to incision.
  Arms: Standard removal technique + lidocaine injection
Device: RemovAid device + lidocaine injection — The RemovAid device incises the skin and grasps the implant for removal. A lidocaine injection will be used prior to incision.
  Arms: RemovAid Device + lidocaine injection

SUMMARY:
This randomized trial will compare different approaches to removing a subdermal contraceptive implant from the upper arm of 225 women in Uganda. The experimental approach is a hand-held device (RemovAid) that incises the skin and grasps the implant for extraction. Safety and efficacy endpoints will be compared to the traditional removal approach (scalpel, forceps, tweezers).

DETAILED DESCRIPTION:
The trial assigns participants to one of three arms: RemovAid+lidocaine patch (n=75), RemovAid+lidocaine injection (n=75) or traditional approach+lidocaine injection(n=75). Complication rates in the different arms will be compared. Efficacy (successful implant removal) will be the secondary comparisons. Finally, pain during removal and duration of removal procedure will be compared. Participants will return to the clinic within 4 weeks of the removal procedure to record the healing process and final interventions (if any).

ELIGIBILITY:
Inclusion Criteria:

* seeking voluntary removal of a one-rod subdermal implant
* willing to sign an informed consent document
* willing to be randomized to the new device vs. standard technique
* willing to follow-up at the study clinic for any subsequent removal-related complications
* willing to have any follow-up complications recorded and shared
* has an implant that is completely and easily palpable
* has an implant that is easily pinched and lifted
* no known allergies to skin preparation products or local anesthetics

Exclusion Criteria:

* Implants that are not easily palpable
* Previous failed implant removal

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Number of women who have post-removal complications - | 4 weeks
  Complications will include unusual level of trauma to the skin (bruising/hematoma), excessive bleeding, use of sutures to repair skin after removal, inability to remove the implant, implant breakage or severing at time of removal, subsequent infection at the removal site, and other complications that may be noted by the investigator
Number of implants that are successfully removed | 0-3 hours
  The number of implants successfully removed i) without breaking the implant and without additional tools (scalpel, tweezers, or forceps), ii) without additional tools, iii) without the additional use of a scalpel.

SECONDARY OUTCOMES:
Participant pain level | 0-3 hours
  Level of pain as recorded on 10cm visual analog scale from 0cm (No Pain) to 10cm (Worse Pain Imaginable) with higher numbers indicating worse outcomes
Duration of removal procedure | 0-3 hours
  Number of minutes and seconds need to remove the implant
Provider feedback on device on whether RemovAid device helped with removal of implant | 0-3 hours
  5-point Likert scale measuring from 1(Strongly Disagree), 2 (Disagree), 3 (Neutral), 4 (Agree), 5 (Strongly Agree) on whether RemovAid device helped with removal of implant with higher scores indicating better outcomes
Provider feedback on device on ways the product helped or hindered implant removal | 0-3 hours
  Text responses on ways the product helped or hindered implant removal

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell-Danielsson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Kawempe Referral Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Results and data will be archived in the Norwegian Social Science Data Services (NSD). Data will be made available after the primary results are published.
Time Frame: Within 24 months after trial completion
Access Criteria: open

REFERENCES:
- [Background] Levine JP, Sinofsky FE, Christ MF; Implanon US Study Group. Assessment of Implanon insertion and removal. Contraception. 2008 Nov;78(5):409-17. doi: 10.1016/j.contraception.2008.06.016. Epub 2008 Sep 18. PMID 18929739
- [Background] Fraser IS. The challenges of location and removal of Implanon contraceptive implants. J Fam Plann Reprod Health Care. 2006 Jul;32(3):151-2. doi: 10.1783/147118906777888459. No abstract available. PMID 16857065
- [Background] Creinin MD, Kaunitz AM, Darney PD, Schwartz L, Hampton T, Gordon K, Rekers H. The US etonogestrel implant mandatory clinical training and active monitoring programs: 6-year experience. Contraception. 2017 Feb;95(2):205-210. doi: 10.1016/j.contraception.2016.07.012. Epub 2016 Jul 21. PMID 27452317
- [Derived] Hubacher D, Byamugisha J, Kakaire O, Nalubwama H, Emtell Iwarsson K, Bratlie M, Chen PL, Gemzell-Danielsson K. Removal of a well-palpable one-rod subdermal contraceptive implant using a dedicated hand-held device or standard technique: a randomized, open-label, non-inferiority trial. Hum Reprod. 2022 Sep 30;37(10):2320-2333. doi: 10.1093/humrep/deac179. PMID 35960174

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT04120337/SAP_000.pdf